CLINICAL TRIAL: NCT02819167
Title: Neuro-anatomical Correlates on Volumetric MRI on the Impact of Brain Reserve and Cognitive Reserve on Ischemic Strokes in Elderly
Brief Title: Brain and Cognitive Reserve
Acronym: BCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0151
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Brain Ischemia
Keywords: ischemic stroke; brain reserve; cognitive reserve; cognitive prognosis
MeSH Terms: conditions — Brain Ischemia; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neurologic and neuropsychological evaluation (Other)
  Interventions: Other: neurologic and neuropsychological evaluation

INTERVENTIONS:
Other: neurologic and neuropsychological evaluation — cognitive prognosis, cognitive reserve, brain volume will be studied on patients with scale, questionnaire, magnetic resonance imaging

SUMMARY:
Ischemic strokes are one of the leading causes of handicap and death in elderly people in France.

Cognitive reserve (CR) is an active model, defined as a function of lifetime intellectual activities and other environmental factors that explain differential susceptibility to functional impairment in the presence of pathology or other neurological insult. CR is estimated using variables for cognitive activity: years of education, professional status, socioeconomic status… Furthermore, brain reverse (BR) is a passive and quantitative model that depend on brain size and other quantitative aspects of the brain that explain differential susceptibility to functional impairment in the presence of pathology.

Firstly, volume and localization of ischemic strokes have a great impact on CR and BR due to brain injury. On the other hand, CR influences the severity and the expression of cognitive diseases.

The investigators realize a prospective study in order to assess the impact of CR and BR on cognitive prognosis after a right middle cerebral artery ischemic stroke in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years old
* right middle cerebral artery ischemic stroke
* hospitalized in neurovascular unit of Pierre Wertheimer hospital between January 2015 to January 2016

Exclusion Criteria:

* Contraindication for MRI
* Hemorrhagic stroke
* Aphasia

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
evaluation of cognitive prognosis | one year post Ischemic stroke
  measure will be performed with the Mattis dementia rating scale

SECONDARY OUTCOMES:
Volume of leucoencephalopathy | one year post Ischemic stroke
  measure will be performed with a MRI
volume of hippocampic | one year post Ischemic stroke
  measure will be performed with a MRI
brain injury | one year post Ischemic stroke
  measure will be performed with a MRI
volume of ischemic stroke | one year post Ischemic stroke
  measure will be performed with a MRI
evaluation of cognitive reserve | one year post Ischemic stroke
  measure will be performed with the Cognitive reserve index questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krolak Salmon, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital des Charpennes, Lyon, France